CLINICAL TRIAL: NCT02029560
Title: Observational Study to Evaluate Effect of Thrupas® Capsule on Cardiovascular System in Patients With Lower Urinary Tract Symptoms Suggestive of Benign Prostatic Hyperplasia
Brief Title: Observational Study to Evaluate Effect of Thrupas® Capsule on Cardiovascular System
Acronym: CV
Status: Completed | Type: Observational
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JWP-SDS-405
Record Dates: First submitted 2013-11-25; First posted 2014-01-08 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate effect on cardiovascular system(blood pressure) when Thrupas® capsule is administered every day for 12 weeks in patients with Lower Urinary Tract Symptoms suggestive of Benign Prostatic Hyperplasia

DETAILED DESCRIPTION:
BPH and hypertension are chronic senile diseases that increase in prevalence with age. It is reported that 25% of men over 60 years old suffer from both BPH and hypertension. Though these two diseases differ in nature, there is a hypothesis advanced from recent studies that for both diseases, increase in sympathetic tone plays an important role in pathophysiology.

As a medical treatment of BPH, α-blockers are widely selected in clinical studies as a first line treatment in patients with LUTS, for its non-invasiveness and superior clinical efficacy [1, 5]. Such α-blockers increases urine flow and decreases residual urine by controlling excitement of the sympathetic nervous system distributed around smooth muscle of prostate and bladder neck. Through this, α-blockers improve conditions of clinical symptoms of patients suffering from LUTS due to BPH, and decrease need for invasive surgery related to BPH, and also have medical action to decrease morbidity rate of secondary complications of BPH such as acute retention of urine, deterioration of renal function, bladder stone and urinary tract infection.

However, in the case of patients who are on hypertension medication, when considering concomitant administration with α-blockers, adverse events such as orthostatic hypotension and dizziness due to drop in blood pressure is most concerned. In this regard, silodosin, as an alpha 1A adrenoceptor antagonist, has been proven have low occurrence of adverse events related to cardiovascular system and have little effect on blood pressure compared to other α-blockers.

Thus, in this study, we aim to see the effect on cardiovascular system(blood pressure) Thrupas® capsule is administered every day for 12 weeks in patients with LUTS suggestive of BPH.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been diagnosed with BPH by digital rectal exam or ultrasonographic findings and meet the following criteria.

1. Male, 50 years or older
2. Patients with a total I-PSS score ≥ 8
3. Patients with a QoL score ≥ 3
4. Patients who voluntarily decided to participate and have filled out consent form

Exclusion Criteria:

1. Patients with an allergy to α-blockers
2. Patients with history of severe arrhythmia, cardiac failure, cardiac infarction, unstable angina, cerebral infarction within 6 months
3. Patients with severe hepatic disorders (hepatic insufficiency, cirrhosis, jaundice, hepatoma)
4. Patients with renal dysfunction
5. Has PSA value ≥ 10ng/ml or has been diagnosed with tumor by biopsy even if PSA value is lower than 10ng/ml,
6. Patients with history of prostate surgery
7. Patients previously administered with 5α-reductase inhibitor within 3 months
8. Patients previously administered with α1-adrenoceptor antagonist within 1 month
9. Patients who are taking the following drugs at the start of study or those who have to take during the 12 weeks of the study: αβ-adrenoceptor antagonist, α-adrenoceptor agonist, anticholinergic (tolterodine, oxybutynin, etc.)
10. Patients with a history of intrapelvic radiation therapy or prostatic hyperthermia

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of study subjects was calculated based on safety end-point which was variable change in SBP measurement before and after the administration of Silodosin. In previous studies, the standard deviation in before and after administration of Silodosin was 12.81. Therefore, this study assumed the standard deviation in before and after administration to be 12.81.
  When the significance level was 0.05, the confidence interval was 1.41 and standard deviation of SBP measurement before and after the administration of Silodocsin was 12.81, the standard sample size will be 318 people and target number of study subject will be 400 as the expected drop rate is 20%.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure (systolic, diastolic) before and after administration | 3 months

SECONDARY OUTCOMES:
Change in IPSS total score before and after administration* | 3 months
Change in QoL score before and after administration | 3 months
Change in IPSS subscore before and after administration | 3 months
Evaluation of BSW after administration | 3 months
Change in Qmax before and after administration | 3 months
Adverse events | 3 months

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Gangam Severance Hospital, Seoul
  - Seoul St. Mary's Hospital of the Catholic University of Korea, Seoul
  - Asan Medical Center, Seoul